CLINICAL TRIAL: NCT05500378
Title: The Effects of a Specific Exercise Program on Subjects With Cervicogenic Headache
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough subjects
Sponsor: Florida Gulf Coast University (Other)
Responsible Party: Principal Investigator, Dr. Rob Sillevis,, Associate Professor, Florida Gulf Coast University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-21
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Cervicogenic Headache
Keywords: Cervicogenic headache; MSK Ultrasound; Obliquus capitis minor; Rectus capitis major; Exercise
MeSH Terms: conditions — Post-Traumatic Headache; Motor Activity

STUDY DESIGN:
Intervention Model Description: One group design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neck extension group (Other): Neck extension group
  Interventions: Other: Head extension and rotation movement

INTERVENTIONS:
Other: Head extension and rotation movement — Active exercise of the head

SUMMARY:
This study explores with the use of MSK Ultrasound imaging if the obliquus capitis minor and the rectus capitis major can be contracted with specific exercises.

DETAILED DESCRIPTION:
This study explores if a subject with the neck in full maximal flexion is able to selective contract the the obliquus capitis minor and the rectus capitis major by head extension and rotation while maintaining the spine position. MSK Ultrasound imaging will be used to measure changes both in length and width.

ELIGIBILITY:
Inclusion Criteria:

* No history of surgery, No current neck pain, Being able to move the neck actively, being able to read English, between ages 18-65

Exclusion Criteria:

* Neck pain, History of surgery, unable to move the head into extension, outside age requirements, unable to read English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
MSK US image | The change in muscle length and diameter will be measured during head movement
  Assessment of change in width and length of target muscles

CONTACTS AND LOCATIONS:
Overall Officials: Rob Sillevis, phD, Principal Investigator — Florida Gulf Coast University
Locations (1):
- Florida Gulf Coast University, Fort Myers, Florida, United States

IPD SHARING:
Plan to Share IPD: No